CLINICAL TRIAL: NCT04759872
Title: Insulin and Muscle Fat Metabolism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unsuccessful enrollment during COVID-19 pandemic.
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Sean Newsom, Associate Professor, Oregon State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-2020-0768
Record Dates: First submitted 2021-02-09; First posted 2021-02-18 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Overweight and Obesity; Insulin Resistance; Metabolic Disease; Mitochondrial Metabolism; Sedentary Lifestyle
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Metabolic Diseases; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be asked to complete 1 screening visit to determine eligibility.
  If participants remain eligible, they will be asked to complete 1 metabolic study visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic Study Visit (Experimental): Participants will complete a study visit for metabolic phenotyping and determination of the impact of hyperinsulinemia on outcomes of interest.
  Interventions: Other: Hyperinsulinemic-euglycemic Clamp

INTERVENTIONS:
Other: Hyperinsulinemic-euglycemic Clamp — Participants will be administered a constant-rate insulin infusion (to induce mild hyperinsulinemia), with an infusion of dextrose to maintain blood glucose concentration (to maintain euglycemia).

SUMMARY:
Our objective in this study is to identify the extent to which insulin drives the accumulation of lipids in skeletal muscle of humans. We will test the hypothesis that 4-hours of mild hyperinsulinemia will result in significant muscle lipid accumulation and that such effects will be similar in lean and overweight/obese humans.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-55 years
* Body mass index (BMI) 18-45 kg/m2
* Sedentary (<1 hour of planned exercise per week)

Exclusion Criteria:

* Regular exercise (>1 hour of planned exercise per week)
* Smoking, tobacco or nicotine use within the last 1-year
* Fasting glucose >126mg/dL
* Hypertension (systolic pressure >140 mmHg or diastolic pressure >90 mmHg)
* Chronic metabolic or cardiovascular health conditions
* Pregnant, nursing, irregular menses or post-menopausal
* Lidocaine allergy
* Certain medications
* Diminished capacity for consent

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Changes in skeletal muscle lipid content during hyperinsulinemia compared with basal resting conditions | Muscle samples will be collected in basal and hyperinsulinemic conditions separated by ~4.5 hours during the metabolic study visit
  Liquid chromatography tandem mass spectrometry (targeted lipidomics) will be used to assess species-level changes in skeletal muscle lipid content in biopsy samples collected before and after the insulin infusion to induce mild hyperinsulinemia.

SECONDARY OUTCOMES:
Changes in skeletal muscle mitochondrial oxidative capacity during hyperinsulinemia compared with basal resting conditions | Muscle samples will be collected in basal and hyperinsulinemic conditions separated by ~4.5 hours during the metabolic study visit
  High-resolution respirometry will be used to assess changes in skeletal muscle mitochondrial oxidative capacity in biopsy samples collected before and after the insulin infusion to induce mild hyperinsulinemia.

CONTACTS AND LOCATIONS:
Overall Officials: Sean A Newsom, Ph.D., Principal Investigator — Oregon State University; Matthew M Robinson, Ph.D., Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No